CLINICAL TRIAL: NCT05021432
Title: Comparison of Virtual Reality And Task Oriented Circuit Training On Gait, Balance and Cognition Among Elderly Population
Brief Title: Virtual Reality And Task Oriented Circuit Training Among Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/00831 Qudsia M
Record Dates: First submitted 2021-08-03; First posted 2021-08-25 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Elderly

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Virtual Reality group will receive video based games training.
  Interventions: Other: Virtual reality training group
- Circuit Training Group (Active Comparator): They will receive Task-oriented Circuit training exercise program
  Interventions: Other: Circuit Training group

INTERVENTIONS:
Other: Virtual reality training group — This group will receive video based games
  Arms: Virtual Reality Group
Other: Circuit Training group — They will receive Task-oriented Circuit training exercise program
  Arms: Circuit Training Group

SUMMARY:
There is a paucity of literature in studying the comparative effects of Virtual Reality and Circuit training in elderly population for fall prevention. This study will also analyze the effects of the comparative intervention on Gait, Balance and Cognition. This will also deduce the impact of Virtual reality and Circuit training on Quality of Life QOL.

DETAILED DESCRIPTION:
As the individual ages, numerous physical and functional alterations occur especially frailty, disturbed body balance, physical and cognitive declines, impaired gait hence leading to falls among the elderly population. Fall is defined as an event in which an individual unintentionally loses balance and inadvertently coming to rest on ground or lower surface. While Balance is the ability to maintain the center of mass on the base of support (BOS) without causing a fall. According to WHO survey, falls are the second leading cause of accidental or unintentional injury deaths worldwide. Approximately 40% of older adults >65years fall at least once a year and 10-20% of these falls results in hospitalizations which leads to poor Quality of Life. Women are more prone for age specific fall rates as compared to men. Cognition is referred to as "The mental action or process of acquiring knowledge and understanding through thought, experience, and the senses". Optimum cognitive levels are important for successful aging and any deficits should be monitored. Altered cognition affects the Activities of Daily living (ADL), causes disabilities and directly impacts the Quality of Life. A study by Ray et al, deduced that Cognitive training significantly increased the Gait speed and improved the Timed up and go test values, hence Cognitive training slows degradation of balance and improves gait while distracted, rendering it a promising approach to falls prevention.

United States Preventive Service Task Force (USPSTF), evaluated that risk of falls increases with age and include multiple factors: Balance and gait deficits, cognitive impairments, medications, frailty, fear of falling, vision and environmental hazard. USPSTF recommends multifactorial interventions to address the balance and fall related issues among elderly. These protocols include improving Balance and gait, improving cognition, environmental alterations, balanced diet and nutrition along with appropriate medications. Adequate exercises helps to improve general body conditioning to overcome the deteriorating effects of aging hence, better Quality of life QOL. Previously it has been reported that a number of specific approaches are useful in improving balance, gait and cognition as compared to general conventional therapies: they include Virtual Reality, Goal oriented training, Task-oriented training, Kinect training and Visual feedback, Motivational interventions with active participations and Focused repetitive training.

As the technological advancement has occurred in recent years, "Virtual Reality" is being incorporated in the PT management sessions to minimize the limitations in the existing interventions and hence improving the deficits. VR training refers to interactive stimulations enabling the user to experience the virtual environment similar to reality by incorporating computer hardware and software. In comparison to home-based exercise plans, VR training enhances motivation by introducing practical gaming element. A Study conducted by on elderly 60-85yrs and they assessed the effects of Wifiit VR games and found that the scores of body Center of pressure-COP movement area (Romberg test) with eyes open and eyes closed improved among experimental group individuals after 8 weeks of trials hence improved Balance. Likewise as reported , VR game exercises improves balance and gait in elderly over 65 yrs of age - increases the step length while average Sway time and Time up and go test TUG both decreased towards normal as compared to conventional Ball exercises.

Task oriented Circuit training CT is a series of systematically devised protocol, which embodies multiple endurance and strength training parameters with moderate and high intensities and sufficient repetitions of functional tasks. As reported that Circuit training improves the partial O2 concentration, Respiratory rate-RR, HR hence overall cardiac endurance and physical functioning. CT also helps in maintenance of functional Quality of life. Several studies have reported that Virtual Reality and Task-oriented circuit training also assists in motor and balance recovery among the stroke and CP. As documented by Lee et al,(13) they compared the effects of VR against CT among the stroke patients and concluded that static balance and Functional reach test outcomes were higher in VR group as compared to CT group hence making Virtual Reality more feasible for balance training. A study concluded that on older adults and deduced that VR training causes improvement in hip muscle strength of the extensors, flexors, adductors, and abductors after 8 weeks along with greater ground reaction force on the backward stepping test (with eyes opened and closed) and the crossover stepping test( with eyes open and closed).

ELIGIBILITY:
Inclusion Criteria:

* • Age between 60-75 years

  * Both Gender
  * In past year-accidental fall history of 1-2 times
  * Be identified as being at medium risk for a fall on the initial medical assessment (Berg balance scale 21- 40/56)
  * Score >19 on SMMSE

Exclusion Criteria:

* • Declared unfit for physical activities following medical assessment.

  * Present with progressive Neurological disease, Vestibular disease or any comorbidity

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Timed up and go test | 8th Weeks
  helps to measure the functional ability and to determine the dynamic balance abilities among the elderly. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling. Change from Baseline balance to 8th Weeks
Dynamic Gait Index | 8th Weeks
  it helps to measure the functional ability and to determine the dynamic balance and gait abilities. its total score is 24. Change from Baseline balance to 8th Weeks

SECONDARY OUTCOMES:
SF-12 scale | 8 Weeks
  The Short Form Health survey questionnaire SF-12 is a preferable instrument for use among the elderly population in order to calculate the Quality of Life.wo summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average. Change from Baseline balance to 8th Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MS, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Pakistan General Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caixeta GC, Dona F, Gazzola JM. Cognitive processing and body balance in elderly subjects with vestibular dysfunction. Braz J Otorhinolaryngol. 2012 Apr;78(2):87-95. doi: 10.1590/S1808-86942012000200014. PMID 22499375
- [Background] Moylan KC, Binder EF. Falls in older adults: risk assessment, management and prevention. Am J Med. 2007 Jun;120(6):493.e1-6. doi: 10.1016/j.amjmed.2006.07.022. PMID 17524747
- [Background] Phu S, Vogrin S, Al Saedi A, Duque G. Balance training using virtual reality improves balance and physical performance in older adults at high risk of falls. Clin Interv Aging. 2019 Aug 28;14:1567-1577. doi: 10.2147/CIA.S220890. eCollection 2019. PMID 31695345
- [Background] de Vries AW, Faber G, Jonkers I, Van Dieen JH, Verschueren SMP. Virtual reality balance training for elderly: Similar skiing games elicit different challenges in balance training. Gait Posture. 2018 Jan;59:111-116. doi: 10.1016/j.gaitpost.2017.10.006. Epub 2017 Oct 5. PMID 29028622
- [Background] Pointer S. Trends in hospitalised injury, Australia. Canberra: Australian Institute of Health and Welfare. 2013.
- [Derived] Ghous M, Masood Q, Nawaz Malik A, Afridi A, Mehmood Q. Comparison of Nonimmersive Virtual Reality and Task-Oriented Circuit Training on Gait, Balance, and Cognition Among Elderly Population: A Single-Blind Randomized Control Trial. Games Health J. 2024 Jun;13(3):164-171. doi: 10.1089/g4h.2022.0205. Epub 2024 Mar 21. PMID 38512706